CLINICAL TRIAL: NCT02309775
Title: Auriculotherapy in Tension-type Headache Due to Temporomandibular Dysfunction - A Randomized Study
Brief Title: Auriculotherapy in Tension-type Headache Due to Temporomandibular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Gabriella de Paula Marcondes Ferreira Leite, Post-graduate student, Federal University of Minas Gerais
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Universidade Federal Alfenas
Record Dates: First submitted 2014-11-18; First posted 2014-12-05 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Auriculotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auriculotherapy Group (Active Comparator): The placement, points according to Souza (1997), will be: Shen Men, Sympathetic, Kidney, Subcortex, Adrenal and Cerebral. The point descriptions are: Shen Men, is located in the vertex of the angle formed by the lower root and the upper root of the antihelix; the Sympathetic is situated in the middle of the lower root below the Helix membrane (located at the lower end of the Lobe); the Kidney point is situated in cymba concha, near its junction with the lower root of the antihelix, in the same line as the Shen Men point; the Subcortex is situated on upward curve towards the apex of the antitragus, on the upper edge of the concha; the Adrenal is located at the apex of the tragus, on its projection towards the concha cava; the Cerebral point is situated above the edge of the antitragus. As sessions will held twice a week for a total of 10 sessions.
  Interventions: Other: Auriculotherapy
- Placebo Grup (Placebo Comparator): The point stimulated will be the Trachea, which is one millimeter in the direction of the auditory meatus. This point does not cause risk to the research participant. As sessions will held twice a week for a total of 10 sessions.

INTERVENTIONS:
Other: Auriculotherapy — First cleaning of the ear is made with 70% alcohol. The seed will be stuck in the ear with an adhesive (Micropore 3M) tape. The placement, points according to Souza (1997), were: Shen Men, Sympathetic, Kidney, Subcortex, Adrenal and Cerebral. As sessions will held twice a week for a total of 10 sessions.
  Arms: Auriculotherapy Group

SUMMARY:
Objectives: Verify the effect of auriculotherapy in patients with tension-type headache resulting from temporomandibular dysfunction.

Design: Randomized clinical study Setting: Randomized Study Participants: The study consist of 38 participants randomized into two groups: an intervention group (n = 18, sample loss = 1) and placebo group (n = 20, sample loss = 6) Interventions: The intervention group will receive treatment with auricular acupuncture in the Shen Men, Kidney, Sympathetic, Subcortex, Adrenal and Cerebral points. The placebo group will receive auriculotherapy in the trachea point.

Main outcome measures: visual analog scale for pain pain (VAS) and surface electromyography (EMG).

DETAILED DESCRIPTION:
This is an experimental clinical trial in which will be selected at the University, 40 students with tension-type headache due to temporomandibular dysfunction. Among the selected subjects will be randomized by blind draw into two groups: intervention group (IG) and placebo group (GII).

The instruments that will be used for the evaluation are the visual analog pain scale, the Survey questionnaire for Temporomandibular Disorders (RDC) 3, and surface electromyography (EMG System of Brazil).

The EMG signals will be collected in the rest position (3 samples) and maximum voluntary isometric contraction (3 collections). The masseter and temporalis muscles bilaterally will be evaluated according to the protocol of Rodrigues.

For treatment of Ear, initially cleaning the pinna is made to be manipulated with 70% alcohol and later will be inserted mustard seed with a tape in the following points: Shenmen, Sympathetic, Kidney, subcortex, Adrenal and Brain second Souza in GI and GII point of the trachea. Such treatment will last 15 minutes each session, being held 2 times a week, alternating the ear to be manipulated over a period of 5 weeks.

For comparison between groups the Mann-Whitney test statistic with Software BioStat 4.0 software will be used. With a significance level (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with tension-type headache due to temporomandibular dysfunction, aged 20 to 30 years, of both sexes

Exclusion Criteria:

* Individuals with migraine type headache, secondary headaches
* Use of medicines more than 10 days per month and any type of acupuncture treatment in the last 12 months

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pattern of muscle contraction (Electromyographic signals of the masseter and temporalis muscles bilaterally.) | one day
  Electromyographic signals of the masseter and temporalis muscles bilaterally.

SECONDARY OUTCOMES:
Pain at the time (Visual analog pain scale) | one week
  Pain at the time will using Visual analog pain scale.